CLINICAL TRIAL: NCT04634695
Title: Assessing the Prevalence and Impact of Dihydropteroate Synthase-431V Mutation on the Protective Efficacy of Intermittent Preventive Treatment During Pregnancy Using Sulphadoxine-pyrimethamine
Brief Title: Assessing to What Extent Dhps-431V Mutation May Influence the Protective Efficacy of IPTp-SP
Acronym: DEEM-FIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Obafemi Awolowo University (Other)
Collaborators: University of Copenhagen (Other); London School of Hygiene and Tropical Medicine (Other); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Sponsor
Other Study IDs: DEEM-FIT
Record Dates: First submitted 2020-11-02; First posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Pregnancy Malaria
Keywords: Antimalarial drug; Sulphadoxine-pyrimethamine; SP-resistance; Malaria in Pregnancy; mutation; Intermittent Preventive treatment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — Whole blood will be collected and DNA will be extracted for malaria parasite genomic analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Malaria in pregnancy (MiP) continues to be a significant public health issue, particularly in sub-Saharan Africa. The coverage of pregnant women with three or more doses of intermittent preventive treatment using sulphadoxine-pyrimethamine (IPTp-SP) is recommended to prevent risks associated with MiP in moderate-to-high transmission settings. Evidence has recently become available supporting the emergence of a novel Pfdhps-431V mutation in Nigeria. This new mutation may further confound the existing SP-resistance; thus, the intended follow-on project aims to assess the influence of Pfdhps-431V mutation on the protective efficacy of SP during pregnancy.

The aims are to detect P. falciparum positivity at delivery and pregnancy outcome in participants who must have received three or more doses of IPTp_SP. We will attempt to check the presence of existing and new Pfdhps/Pfdhfr mutations in the samples positive for P. falciparum using a quantitative PCR (qPCR). The prevalence of novel Pfdhps-431V mutant and other Pfdhps/Pfdhfr resistance alleles among the study population will be estimated. The significance of the resistance genes on the efficacy of SP will be described by looking at its associations with the reported IPTp use, P. falciparum infection, maternal anaemia, low birth weight, and preterm delivery.

DETAILED DESCRIPTION:
Malaria in pregnancy (MiP) is considered a major public health issue with substantial risks for mothers and their babies. Intermittent preventive treatment in pregnancy using sulphadoxine-pyrimethamine (IPTp-SP) is adopted as a part of antenatal care (ANC) to prevent malaria and reduce the risk associated with MiP. However, SP-resistance is increasing with the emergence of Plasmodium falciparum dihydropteroate synthase (Pfdhps) and P. falciparum dihydrofolate reductase (Pfdhfr) resistant genes challenging the benefits and effectiveness of IPTp-SP. Still, evidence has become available supporting the emergence of a novel Pfdhps-I431V mutation. The I431V mutation is found only in West and Central African countries, however, its impact on SP resistance has not been evaluated. We are hypothesizing that the new mutation may confound the existing SP-resistance resulting in an apparent reduction in the protective effect of SP during pregnancy within the region.

The study will recruit adult pregnant women and will assess the presence of malaria infection at delivery. The study will seek new mutations in vivo using full sequencing. This molecular tool will also be used to look at the prevalence of novel Pfdhps-431V mutation among pregnant women undergoing monthly IPTp-SP. Attempts will be made to re-evaluate the prevalence of other Pfdhps and Pfdhfr resistance alleles among the study population. The significance of the resistance genes on the protective efficacy of SP will be described.

The present study is an observational study to be conducted among all booked pregnant women. The pregnant women must have received at least three therapeutic doses of sulphadoxine-pyrimethamine as part of routine antenatal care (ANC) before delivery. sion and Pregnant women who consented to participate will be tested for the presence of malaria parasite during the third trimester and at delivery. 80-100 µL blood samples will be saved as dried blood spot on Whatman® filter paper from the individual with P. falciparum malaria positivity Antenatal care (ANC) contact schedule with proposed timelines for implementation of malaria in pregnancy interventions designed by WHO will be followed in enrolling subjects from 26 weeks of pregnancy. The study will be conducted at the antenatal

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at 26 weeks of pregnancy who aged ≥ 18 years; Must have commenced IPTp-SP and intended to receive three or more therapeutic doses of SP before delivery; Readiness to give informed consent and comply with the study protocol.

Exclusion Criteria:

* Pregnant women during their first trimester as SP is not recommended during the first trimester; Severe or complicated malaria as the subject will require additional treatment and consideration; Presence of underlying chronic or severe diseases (e.g., cardiac, renal or hepatic diseases, HIV/AIDS); Individuals who are receiving co-trimoxazole for another disease condition (as SP is not usually recommended): Inability to swallow oral medication because of persistent nausea and vomiting

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Antenatal care (ANC) contact schedule with proposed timelines for implementation of malaria in pregnancy interventions designed by WHO(16) will be followed in recruiting subjects from 26 weeks of pregnancy. The study will be conducted at the antenatal clinics of Obafemi Awolowo University Teaching Hospitals complex, Ile-Ife
Sampling Method: Non-Probability Sample
Enrollment: 288 (Estimated)
Dates: Start 2020-08-10 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Malaria infection at the time of delivery | May 2021
  P. falciparum malaria positivity will be confirmed using microscopy
Dhps-431V mutation | May 2021
  Point mutation at codon dhps-I431V will be carried out

SECONDARY OUTCOMES:
Average maternal haematocrit | May 2021
  Maternal haematocrit will be carried out to confirm whether the mother is anaemic or not
Birth weight of babies | May 2021
  Birth weight of babies
Prevalence of placental malaria | May 2021
  Prevalence of placental malaria

CONTACTS AND LOCATIONS:
Overall Officials: Adebanjo Adegbola, PhD, Principal Investigator — Obafemi Awolowo University
Locations (2):
- Nigeria (2):
  - Obafemi Awolowo University Teaching Hospital, Ile-Ife, Osun State
  - State Specialist Hospital, Asubiaro, Osogbo, Osun State

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van Eijk AM, Larsen DA, Kayentao K, Koshy G, Slaughter DEC, Roper C, Okell LC, Desai M, Gutman J, Khairallah C, Rogerson SJ, Hopkins Sibley C, Meshnick SR, Taylor SM, Ter Kuile FO. Effect of Plasmodium falciparum sulfadoxine-pyrimethamine resistance on the effectiveness of intermittent preventive therapy for malaria in pregnancy in Africa: a systematic review and meta-analysis. Lancet Infect Dis. 2019 May;19(5):546-556. doi: 10.1016/S1473-3099(18)30732-1. Epub 2019 Mar 25. PMID 30922818
- [Result] Oguike MC, Falade CO, Shu E, Enato IG, Watila I, Baba ES, Bruce J, Webster J, Hamade P, Meek S, Chandramohan D, Sutherland CJ, Warhurst D, Roper C. Molecular determinants of sulfadoxine-pyrimethamine resistance in Plasmodium falciparum in Nigeria and the regional emergence of dhps 431V. Int J Parasitol Drugs Drug Resist. 2016 Dec;6(3):220-229. doi: 10.1016/j.ijpddr.2016.08.004. Epub 2016 Sep 29. PMID 27821281
- [Result] Alifrangis M, Nag S, Schousboe ML, Ishengoma D, Lusingu J, Pota H, Kavishe RA, Pearce R, Ord R, Lynch C, Dejene S, Cox J, Rwakimari J, Minja DT, Lemnge MM, Roper C. Independent origin of plasmodium falciparum antifolate super-resistance, Uganda, Tanzania, and Ethiopia. Emerg Infect Dis. 2014 Aug;20(8):1280-6. doi: 10.3201/eid2008.131897. PMID 25061906